CLINICAL TRIAL: NCT04585178
Title: Detection of Postoperative Complications and Particularly Hemodynamic Ones Through Continuous Monitoring Using the Biobeat Patch
Brief Title: Screening for Postoperative Vital Signs Abnormalities, and Particularly Hemodynamic Ones, by Continuous Monitoring Using the Biobeat Patch
Acronym: Biobeat-Postop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020_0050
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Surgery--Complications
Keywords: surgery; vital signs; continuous monitoring

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biobeat patch (Experimental): Patients will be asked to keep Biobeat patch during 72 hours after their surgery.
  Interventions: Device: Biobeat patch

INTERVENTIONS:
Device: Biobeat patch — The Biobeat device (BB-613WP) is a class IIa medical device and is a non-invasive patch used for monitoring vital signs in clinical and non-clinical settings. The sensor continuously records the photoplethysmographic waveform that allows the calculation of several physiological parameters: heart rate (HR), SPO2, systolic blood pressure (SBP) and change in SBP, diastolic blood pressure (DBP) and change in DBP, stroke volume (SV), cardiac output (CO), cardiac index (CI), systemic vascular resistance (SVR), and respiration rate (RR).
  Translated with www.DeepL.com/Translator (free version)

SUMMARY:
Brief Summary: Post-operative morbidity remains a reality as shown by the International Surgical Outcomes Study published in 2016 and 2019 and by several recent publications which focus mainly on hypotension and cardio-vascular complications. Other complications, such as respiratory depression, are less often studied. The hypothesis is that this connected patch could be used in surgical departments to detect a postoperative complication.

Biobeat Technologies Ltd has developed a sensor which continuously records the photoplethysmographic waveform and allows the calculation of several physiological parameters: heart rate (HR), oxygen saturation (SpO2), systolic blood pressure (SBP), diastolic blood pressure (DBP), stroke volume (SV), cardiac output (CO), cardiac index (CI), systemic vascular resistance (SVR), respiratory rate (RR), and temperature.

The objective of this study is the quantification of hemodynamic, respiratory and temperature abnormalities detected by routine monitoring (routine nursing follow-up) and continuous monitoring by the Biobeat patch during the first 72 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient undergoing major digestive, gynecological, orthopedic or urological surgery (expected duration of surgery greater than 2 hours).
* Predictable postoperative hospitalization duration ≥ 2 nights
* Patient with a Health Insurance plan
* Not having opposed participation in the research

Exclusion Criteria:

* Patient with significant deformity, swelling, irritation or with localized infection, ulceration or skin lesions on the torso
* Patient with a subcutaneous electronic pacemaker implant.
* Patient with a CT or MRI scan already scheduled for the first three days postoperatively
* Patient suffering from tremors or convulsions
* Patient with a torso tattoo
* Patient with significant chest hairiness
* Patient with a known allergy to metals, plastics and silicone
* Patient deprived of liberty or under guardianship
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a hemodynamic abnormality using the data obtained using the Biobeat patch. | 72 hours
  A hemodynamic abnormality is defined as an mean Blood Pressure (MBP) < 60 mmHg

SECONDARY OUTCOMES:
Proportion of patients with hypotension detected by the routine nursing follow-up. | 72 hours
  A hemodynamic abnormality is defined as:
  * An MBP < 70 mmHg
  * or an MBP < 65 mmHg
  * or an MBP < 80% of the value measured during the preanesthetic consultation
  * or an MBP < 70% of the value measured during the preanesthetic consultation
  * or an MBP < 80% of the value measured in the OR before the induction of anesthesia
  * or an MBP < 70% of the MBP measured in the OR before the induction of anesthesia
  * or an MBP > 100 mmHg
  * or an MBP > 110 mmHg
  * or an MBP > 120 mmHg
  * or an MBP > 130 mmHg
  * or an MBP > 120% of the MBP measured during the preanesthetic consultation
  * or an MBP > 130% of the MBP measured during the preanesthetic consultation
  * or an MBP > 120% of the MBP measured in the OR before induction of anesthesia
  * or an MBP > 130% of the MBP measured in the OR before induction of anesthesia
  * or a heart rate < 40/min
  * or a heart rate > 100/min
  * or a rhythm disorder
Proportion of patients with a postoperative respiratory abnormality using the data obtained using the Biobeat patch. | 72 hours
  A postoperative respiratory abnormality is defined as:
  * a breathing rate < 8/min
  * or a breathing rate > 20/min
  * or arterial oxygen saturation < 95%
  * or arterial oxygen saturation ≤ 92%
  * or arterial oxygen saturation ≤ 90%
  * or arterial oxygen saturation ≤ 85%
Proportion of patients with a postoperative respiratory abnormality detected by the routine nursing follow-up. | 72 hours
  A postoperative respiratory abnormality is defined as:
  * a breathing rate < 8/min
  * or a breathing rate > 20/min
  * or arterial oxygen saturation < 95%
  * or arterial oxygen saturation ≤ 92%
  * or arterial oxygen saturation ≤ 90%
  * or arterial oxygen saturation ≤ 85%
Proportion of patients with a temperature abnormality using the data obtained using the Biobeat patch. | 72 hours
  A temperature abnormality is defined as:
  * a temperature ≤ 36.8 °C
  * or a temperature ≥ 38°C
  * or a temperature ≥ 39°C
Quantify and compare the frequency of temperature abnormality detected by the routine nursing follow-up. | 72 hours
  temperature abnormality is defined as:
  * a temperature ≤ 36.8 °C
  * or a temperature ≥ 38°C
  * or a temperature ≥ 39°C
Concerning the Biobeat patch, frequency of artifacts or of absence of data | 72 hours
  An artefact is defined as
  * a value that is > 50% different from the previous value, unless it is followed by a value equal to ± 25%;
  * or a value that is outside the physiologically plausible range (heart rate < 5 or > 250 bpm, systolic blood pressure < 20 mm Hg or > 300 mm Hg or lower than diastolic pressure plus 5 mm Hg, diastolic blood pressure < 5 mm Hg or > 225 mm Hg, change in SpO2 ≥ 8% between two consecutive measurements, breathing rate < 3 or > 125 breaths per minute, change in skin temperature ≥ 1° between two consecutive measurements).
Collection of postoperative complications that occurred during the monitoring period | 72 hours
  A postoperative complication will be classified according to the classification of Dindo and Clavien (Dindo, Demartines et al. 2004).
Evaluation of patients' tolerance to wearing the Biobeat device | 72 hours
  4- point Likert scale (from 0 = intolerable to 4 = no problem at all)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Paternot, Dr, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Groupe hospitalier Paris Saint-Joseph, Paris
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Dryad Repository

REFERENCES:
- [Background] Liem VGB, Hoeks SE, Mol KHJM, Potters JW, Grune F, Stolker RJ, van Lier F. Postoperative Hypotension after Noncardiac Surgery and the Association with Myocardial Injury. Anesthesiology. 2020 Sep;133(3):510-522. doi: 10.1097/ALN.0000000000003368. PMID 32487822
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] International Surgical Outcomes Study (ISOS) group. Prospective observational cohort study on grading the severity of postoperative complications in global surgery research. Br J Surg. 2019 Jan;106(2):e73-e80. doi: 10.1002/bjs.11025. PMID 30620066
- [Background] Turan A, Chang C, Cohen B, Saasouh W, Essber H, Yang D, Ma C, Hovsepyan K, Khanna AK, Vitale J, Shah A, Ruetzler K, Maheshwari K, Sessler DI. Incidence, Severity, and Detection of Blood Pressure Perturbations after Abdominal Surgery: A Prospective Blinded Observational Study. Anesthesiology. 2019 Apr;130(4):550-559. doi: 10.1097/ALN.0000000000002626. PMID 30875354
- [Derived] Paternot A, Aegerter P, Martin A, Ouattara J, Ma S, Adjavon S, Trillat B, Alfonsi P, Fischler M, Le Guen M. Screening for postoperative vital signs abnormalities, and particularly hemodynamic ones, by continuous monitoring: protocol for the Biobeat-Postop cohort study. F1000Res. 2021 Jul 21;10:622. doi: 10.12688/f1000research.54781.2. eCollection 2021. PMID 34754421